CLINICAL TRIAL: NCT02145273
Title: Healthy Moms-Healthy Kids: Reducing Maternal Depression for Better Outcomes in Head Start Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Ferol Mennen, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 90YR0074-01-00; 90YR0074-01 (NIH)
Record Dates: First submitted 2014-05-19; First posted 2014-05-22 (Estimated); Last update posted 2019-06-11 (Actual); Status verified 2017-04

CONDITIONS: Maternal Depression; Parenting Behavior; Health; Interpersonal Relationships; Goal Directed Behavior; Child Behavior; Child School Readiness
Keywords: Maternal Depression; Interpersonal Psychotherapy; School Readiness
MeSH Terms: conditions — Child Behavior | interventions — Interpersonal Psychotherapy

STUDY DESIGN:
Intervention Model Description: There are 3 conditions that will be followed for up to 2 years: control, intervention and comparison. Randomization is by site. Half the sites are control half are intervention. all possible subjects are screened for depression. if the subject is depressed they are invited in to control or intervention based on site, all non depressed subjects are invited into the comparison.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intervention (Experimental): Subjects screen positive for depression and are offered a group Therapy intervention for depression: Interpersonal Psychotherapy for Depression Group.
  Interventions: Behavioral: Interpersonal Psychotherapy for Depression -Group
- Control (No Intervention): Subjects screen positive for depression and are offered Treatment as usual: External referral.
- comparison (No Intervention): Subjects screen negative for depression: no referral or intervention.

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy for Depression -Group
  Arms: Intervention

SUMMARY:
Maternal depression is a pervasive problem that disproportionately affects low-income mothers. The effects of depression on mothers and their parenting result in many negative outcomes for children, particularly in terms of school readiness. The proposed research will build on a successful partnership between the University of Southern California School of Social Work (USC) and Children's Institute, Inc. (CII) to implement and evaluate an evidence-based intervention, interpersonal psychotherapy for group (IPT-G), for Head Start mothers with depression or dysphoric mood with the goal of reducing their depression and promoting positive changes for both mothers and children. The objectives of the study are: (1) adapt IPT-G for a Head Start population of mothers with depression; (2) implement IPT-G via a randomized controlled trial in Head Start centers in Los Angeles County operated by CII; (3) evaluate the effects of the intervention on maternal depression, parenting behaviors, goal-directed behavior, interpersonal relationships, physical health, and child behavior and school readiness; and (4) develop a manual for use of the intervention in Head Start and disseminate findings nationally. The study will feature 2 groups of 60 mothers each, randomized by Head Start site; one will receive the intervention and the other services as usual. Outcomes for both mothers and children will be tracked for 2 years after the intervention, allowing for the evaluation of short- and long-term effects. The intervention will be delivered by Head Start mental health workers under the supervision of Scott Stuart, a national trainer of the intervention. This intervention has the potential to be a low-cost, high-impact intervention that can be replicated to other Head Start sites across the country to improve the lives of Head Start children and families.

ELIGIBILITY:
Inclusion Criteria:

* Mothers of children in Head Start with scores on screening measure that are in depressed or possibly depressed range to be assigned to intervention or TAU. Also will have additional control group of non depressed mothers

Exclusion Criteria:

* Not able to function in group environment

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2014-09; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory | At entry, completion of intervention, and every 6 months for 2 years

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Children's Institute, Inc., Los Angeles, California
  - University of Southern California School of Social Work, Los Angeles, California